CLINICAL TRIAL: NCT02351362
Title: A Pilot Study of a Voucher Incentive System for Improving Retention in Postpartum HIV Care in South Africa
Brief Title: A Pilot Voucher Incentive for Improving Retention in Postpartum HIV Care in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Vanderbilt University (Other); University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Matthew Fox, Associate Professor, Boston University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-33546
Record Dates: First submitted 2015-01-22; First posted 2015-01-30 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: HIV
Keywords: Retention; Attrition; Incentive; Pregnant women
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incentive Group (Experimental): A one-time supermarket voucher of R50 (about $5.00) for participants who return for at least one postpartum visit at the study clinic within 10 weeks of delivery
  Interventions: Behavioral: Incentive Group
- Control Group (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Incentive Group — A one-time supermarket voucher of R50 (about $5.00) for participants who return for at least one postpartum visit at the study clinic within 10 weeks of delivery
  Arms: Incentive Group

SUMMARY:
Given there is substantial loss to follow-up soon after delivery among HIV-positive pregnant women in South Africa, we will conduct a pilot study of an innovative approach to improve retention in care targeted to this specific population at high risk of drop-out. The problem of poor retention in care is well documented, but interventions to address the issue are lacking. In order to design an effective intervention that will be tested in a future randomized controlled trial, we will first complete preliminary research via a pilot study in order to determine the feasibility and acceptability of an incentive program (i.e., a supermarket voucher) to reduce loss to follow-up among HIV-positive women after delivery.

The primary objective of this study is to determine the feasibility of a voucher incentive intervention aimed at improving retention in postpartum HIV care

Secondary objectives include: a) to determine the efficacy of the intervention at increasing postpartum retention; b) to determine the acceptability of the intervention in terms of women's preferences for the intervention compared to other possible interventions; c) to assess differences in patient retention among women newly diagnosed with HIV vs. those who knew their HIV-positive status before pregnancy; and d) to assess differences in patient retention among women who initiated ART during pregnancy vs. those who were on ART before becoming pregnant.

We will enroll up to 200 adult (≥18 years), pregnant, HIV-positive women attending antenatal care who have not previously enrolled in the study at Hikhensile Clinic, Johannesburg, South Africa. The study will be a prospective intervention cohort study with historical controls. Intervention subjects will receive a one-time supermarket voucher of R50 (about $5.00) for participants who return for at least one postpartum visit at the study clinic within 10 weeks of delivery.

DETAILED DESCRIPTION:
STUDY DESIGN

This is a prospective intervention cohort study with historical controls. Since this is pilot study to inform a future intervention, up to 200 participants will be enrolled total: up to 100 to receive the intervention and up to 100 historical controls extracted from electronic clinic records. We are using historical controls because we don't feel it is appropriate to randomize vouchers at a site as this will likely cause ill will in the clinic and the clinic was not willing to do this. We also do not have the resources to get data from a second clinic and we felt that given this was a pilot study we would likely increase confounding if we went to another clinic for a comparison group. While the procedure is changing at the clinic to move to Option B+, we do not anticipate being able to begin the actual intervention until late February or March. This will allow for a sufficient number of historical controls to accrue under option B+ to use as a relevant control group. No patient matching will occur.

STUDY SITE Hikhensile Clinic is a primary health care clinic in Region A of Johannesburg, South Africa, operated by the City of Johannesburg Department of Health. Hikhensile primarily serves clients living in Ivory Park (Ward 77) in Midrand.

Hikhensile Clinic offers antenatal and postnatal care, HIV testing and treatment on-site, as well as other primary care services. HIV care is integrated with antenatal care for pregnant women, with assessment for and initiation of ART occurring within antenatal care. HIV testing occurs during a woman's first antenatal visit and, per national guidelines, all pregnant women will be initiated on lifelong antiretroviral therapy (Option B+) as of in January 2015. Hikhensile does not perform deliveries, so all women who receive antenatal care at Hikhensile are designated to deliver at Tembisa Hospital and Ethafeni Hospital. The hospitals do not routinely report delivery information back to Hikhensile. Following delivery, patients return for postnatal care and HIV treatment services at Hikhensile for 10 weeks and then resume general adult care, all within the same facility and using the same clinic file. Mothers and infants make three postnatal care visits together: 3-7 days after delivery; six weeks after delivery for an infant polymerase chain reaction HIV test to determine the HIV status of the baby; and 10 weeks after delivery for infant HIV results.

STUDY POPULATION The study population will consist of up to 200 HIV-positive pregnant women. Up to 100 will be recruited consecutively and enrolled prospectively during routine antenatal care at Hikhensile Clinic in Johannesburg, South Africa. Patient records for up to 100 HIV-positive pregnant women from Hikhensile will be extracted to serve as the historical control group for comparison.

At the enrollment visit, the following procedures will occur:

1. Pregnant women will be recruited and screened for eligibility for the study by study staff.
2. Women who provide informed consent for participation will be enrolled into the study.
3. The questionnaire (attached in the Appendix) will be administered by trained study staff. The questionnaire is designed to elicit information that is not already collected routinely, including questions related to demographic information, attitudes about the study, and behavioral and socio-economic factors that may influence retention in care. The questionnaire will take about 30-45 minutes to administer.
4. Patients will be reminded that we will also access their medical records to collect information about their medical history and that we may do so up to one year after enrollment to see if their health changes in any way.
5. Study staff will explain how the intervention works, reminding the patient that they must return to the clinic within 10 weeks of delivering their baby to receive the voucher.
6. Staff will also remind the participant that the voucher is a one-time incentive, they will not receive any additional incentives after the initial voucher. They will also be reminded they will not receive the voucher if they return later than 10 weeks after delivery.

Follow-up activities at the first postpartum visit (within 10 weeks of delivery)

1. At the first postpartum visit, it is standard procedure to record the date and details of delivery. If the participant returns to the study clinic within 10 weeks of delivery of the baby, study staff will provide the participant with a R50 supermarket voucher for returning to the clinic. She will need to sign a form that states that she received the form and understands that she will not receive another voucher from the study team or the clinic staff. To receive the voucher a woman must return within 10 weeks of the estimated delivery date as women are supposed to receive 10 weeks of postnatal care at the clinic before transferring to adult HIV care. We will extend the data collection to 14 weeks to see if any women return in the 4 weeks after the intervention period ends. These women will not receive a voucher.

   Follow-up activities approximately 14 weeks after delivery
2. Clinical records will be assessed for all participants a minimum of one month following the scheduled 10-week postpartum visit. If the participant did not return within 14 weeks of delivery, she will be considered to have completed no postpartum visits.

ELIGIBILITY:
Inclusion Criteria:

Adult (≥18 years of age)

* HIV-positive at the time of enrollment
* Pregnant
* Initiating ART on day of enrollment, or already initiated on ART
* Willing and able to provide written informed consent for study participation and data collection
* Able to speak and understand spoken English
* Must possess a working cell phone during the enrollment visit
* Not previously enrolled in the study

Exclusion criteria:

- Patient requests to be transfered to non-study site for HIV care and treatment on day of recruitment/enrollment

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of participants who receive a voucher. | 10 weeks
  Defined as each participant who qualifies for a voucher successfully receiving the voucher via electronic transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Fox, DSc, Principal Investigator — Boston University
Locations (1):
- HIV Clinic, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Undecided